CLINICAL TRIAL: NCT04149340
Title: Comparison of Two Sedation Versus Placebo Techniques on the Patient's Intraoperative Comfort During Cataract Surgery Under Local Anesthesia
Brief Title: Comparison of Two Sedation Versus Placebo Techniques During Cataract Surgery Under Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANESCATARACT
Record Dates: First submitted 2019-10-17; First posted 2019-11-04 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Sedation; Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sufentanil sedation (Other): 3 microgram of Sufentanil IV
  Interventions: Drug: Cataract surgery
- Placebo sedation (Placebo Comparator): 1 ml de NaCl 0,9%
  Interventions: Drug: Cataract surgery
- Multimodal sedation (Other): Clonidine, sufantil, midazolam, dihydrobenzperidol, ketamine
  Interventions: Drug: Cataract surgery

INTERVENTIONS:
Drug: Cataract surgery — Patient's satisfaction and surgeon's satisfaction was assessed by four Lickert's scales, ranging from one to four. hemodynamic parameters before incision, 10 min post-incision and at the end of the surgery

SUMMARY:
Check the sedation conditions during topic cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Topic cataract surgery

Exclusion Criteria:

* NA

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction: four Lickert's scales | During cataract surgery
  The patient's satisfaction was assessed by four Lickert's scales, ranging from one (worse outcome )to four (better outcome)

SECONDARY OUTCOMES:
Surgeon's satisfaction: four Lickert's scales | During cataract surgery
  The surgeons's satisfaction was assessed by four Lickert's scales, ranging from one (worse outcome )to four (better outcome)
hemodynamic parameters | Durinf cataract surgery
  The hemodynamic parameters was rated before incision, 10min after incision and at the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, University Hospital, Liège, Belgium